CLINICAL TRIAL: NCT05697796
Title: Comparison of Post-operative Lower Urinary Tract Symptoms After Sacrospinous Ligament Fixation or Extraperitoneal High Uterosacral Ligament Suspension for Patients With Pelvic Organ Prolapse
Brief Title: Comparison of Post-operative Symptoms After Two Surgeries for Patients With Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Xiuli, Department director, professor, Peking University People's Hospital
Other Study IDs: PKUPH8
Record Dates: First submitted 2022-12-24; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients had pelvic organ prolapse who undergone Sacrospinal ligament fixation
  Interventions: Procedure: Two different surgical methods
- patients had pelvic organ prolapse who undergone Extraperitoneal high sacral ligament suspension
  Interventions: Procedure: Two different surgical methods

INTERVENTIONS:
Procedure: Two different surgical methods — SSLF：sacrospinal ligament fixation EHUS：Extraperitoneal high sacral ligament suspension

SUMMARY:
Collect and review the patients who underwent surgical treatment due to pelvic floor organ prolapse from 2020 to 2021, make statistics on their postoperative questionnaire data, and evaluate the clinical effects of different surgical methods

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years;

  * Because pelvic organ prolapse in our hospital, we performed extraperitoneal high sacral ligament suspension or sacrospinal ligament fixation; ③ Those who have no surgical contraindication and can tolerate surgery and anesthesia.

Exclusion Criteria:

* Those who cannot tolerate surgery and anesthesia; ② Patients receiving other tip suspension techniques.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients had pelvic organ prolapse receiving two specific surgical methods
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
changes in POP-Q score at different time nodes | pre-operation and post-operation(1month, 3 months and 6 months )
  Gynecological examination

SECONDARY OUTCOMES:
UDI-6 scores at different time nodes | pre-operation and post-operation(1month, 3 months and 6 months )
  Questionnaires on lower urinary tract symptoms and quality of life
PFDI-20 scores at different time nodes | pre-operation and post-operation(1month, 3 months and 6 months )
  Questionnaires on lower urinary tract symptoms and quality of life
OABss scores at different time nodes | pre-operation and post-operation(1month, 3 months and 6 months )
  Questionnaires on lower urinary tract symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- The Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes